CLINICAL TRIAL: NCT02341131
Title: BDNF as a Potential Biomarker for Cognitive Remediation Therapy in Schizophrenia
Brief Title: Cognitive Remediation Therapy in Schizophrenia: Effects on BDNF Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Rafael Penades, Ph.D., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 11/01958
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive Remediation; BDNF
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training; Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Remediation Therapy (Experimental): Cognitive Remediation Therapy -Frontal/Executive Program (Delahunty)- (Wykes & Reeder, 2005)
  Interventions: Behavioral: Cognitive Remediation Therapy
- Psychoeducation (Active Comparator): Symptom Management Module from the University of California. Liberman & Kopelowicz (1995)
  Interventions: Behavioral: Psychoeducation
- Healthy Controls (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — The program has a duration of 40 sessions (one hour of duration), with two sessions for week during four months. It is carried out individually and utilizes paper and pencil tasks. The main technique utilized is the scaffolding (to provide strategies when the patient cannot carry out the task and to withdraw him when he is yet able of doing it alone) in a context of learning without errors.
  Other Names: Cognitive rehabilitation, cognitive training
  Arms: Cognitive Remediation Therapy
Behavioral: Psychoeducation — The program has a duration of 40 sessions (one hour of duration), with two sessions for week during four months. It is carried out individually and utilizes teaching information and coping skills and neuropsychological issues are not addressed.
  Other Names: Coping strategies, skills training
  Arms: Psychoeducation

SUMMARY:
The main objective of the study is to analyse the role of a neurotrophic factor (BDNF) as a putative biological marker of the cognitive recovery in schizophrenia following a Cognitive Remediation Therapy (CRT). Additionally, the role as outcome predictors of BDNF serum levels and the Val66met polymorphism and data from functional and structural neuroimaging will be studied.

DETAILED DESCRIPTION:
Forty patients with schizophrenia disorder and twenty healthy volunteers will be recruited. Patients will be randomly allocated either the experimental group, undergoing an individual CRT for 40 hours during 16 weeks, or the control group following a psycho-educational intervention without any neurocognitive work, both lasting the same amount of hours and period of time. Blood samples will be obtained from participants in four moments: before treatment, at week 4, at week 16, and at 32 week follow-up. In addition, repeated measurements will be obtained with a neurocognitive battery based on the MATRICS consensus battery and the Positive And Negative Syndromes Scale (PANSS). Assessments will be conducted by trained personnel who will remain blind to the group assignment. A factorial model will be performed conducting a repeated measures analysis of covariance (ANCOVA) to study the effects of CRT on the levels of BDNF, neurocognition, symptoms and social functioning, adding the necessary co-variants. Finally, a linear regression model to determine the predictive role of serum levels of BDNF and data from functional and structural neuroimaging on the effects of CRT will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV-TR and confirmed by the semi-structured interview (SCID) for the axis 1.
* Presence of cognitive deficit confirmed by the neuropsychological battery
* Stable symptomatology at least during the last six months and the estimation of not modifying pharmacological antipsychotic treatment.

Exclusion Criteria:

* Presence of organic-cerebral affectation due to neurological or traumatic conditions
* Abuse of psychotropic substances
* Presence of other psychiatric symptomatology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
BDNF (change from baseline serum BDNF levels) | Baseline, 1 month and 4 months
  Change Measurements of serum BDNF levels will be carried out by personnel blind to subjects' group assignment. Platelet and serum samples will be diluted with diluent included in the R&D Human BDNF Quantikine Enzym Linked Immunosorbent Assay (ELISA) kit (Yasuhito et al. 1987).

SECONDARY OUTCOMES:
Symptoms (Change from baseline in Positive and Negative Syndrome Scale (PANSS) scores) | Baseline and 4 months
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) scores at time 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Penadés, Ph.D., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Penades R, Segura B, Inguanzo A, Garcia-Rizo C, Catalan R, Masana G, Bernardo M, Junque C. Cognitive remediation and brain connectivity: A resting-state fMRI study in patients with schizophrenia. Psychiatry Res Neuroimaging. 2020 Sep 30;303:111140. doi: 10.1016/j.pscychresns.2020.111140. Epub 2020 Jul 15. PMID 32693320